CLINICAL TRIAL: NCT02624531
Title: Prospective Study of Fertility-sparing Treatment Strategy in Patients With Early Cervical Cancer(SYSUGO-005/CSEM009)
Acronym: SYSUGO-005
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Pro., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-070
Record Dates: First submitted 2015-11-09; First posted 2015-12-08 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Cervical Cancer
Keywords: NACT; Cervical cancer; Fertility sparing; Pregnancy; Treatment Strategy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — taxane; Cisplatin; Conization; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fertility-sparing surgery (Other): NACT with Taxane combined with cisplatin and Fertility-sparing Treatment Strategy
  Interventions: Drug: Taxane; Procedure: radical trachelectomy

INTERVENTIONS:
Drug: Taxane — NACT and Fertility-sparing Treatment Strategy
  Other Names: cisplatin
Procedure: radical trachelectomy — NACT and Fertility-sparing Treatment Strategy
  Other Names: simple trachelectomy; conization; sentinel node biopsy

SUMMARY:
Patients with cervical cancer staging IB1-IIA2 desiring keeping their fertility function will be recruited. Before treatment, MRI scanning will be used to exclude retroperitoneal lymph node metastasis, involvement of lower part of uterus and endometrial carcinoma.If there is no macroscopic tumor and no obvious disease in MRI,simple trachelectomy (ST) + sentinel lymph node biopsy (SLNB) / retroperitoneal lymph node dissection(RPLND) will be performed. Otherwise,two to three cycles of neoadjuvant chemotherapy (NACT) will be administrated and then different fertility-sparing surgery(conization,ST or radical trachelectomy(RT) + SLNB/RPLND) will be employed depending on the tumor size.

DETAILED DESCRIPTION:
The age of patients who are diagnosed with cervical cancer has decreased, resulting in a trend of increasingly younger patients who seek to preserve their fertility. Therefore, a less radical approach that aims to preserve the potential for fertility during the treatment of cervical carcinoma is crucial. Herein, the investigators devote to exploring optimal fertility-sparing treatment strategy in Patients With cervical cancer.

In this study, patients with cervical cancer staging IB1-IIA2 desiring keeping their fertility function will be recruited. Before treatment, MRI scanning will be used to exclude retroperitoneal lymph node metastasis, involvement of lower part of uterus and endometrial carcinoma.

All lymph nodes and margin should be pathologic reviewed during the surgery. Fertility-sparing surgery should be abandoned if positive lymph node is found.

If there is no macroscopic tumor and no obvious disease in MRI, ST+ SLNB/RPLND will be performed. Otherwise, two or three cycles of NACT will be administrated and then chemotherapy response will be assessed with physical examination and MRI scanning.

If there is no obvious residual disease after NACT, the colposcopy will be used to search for the suspicious disease in the cervix and on the vaginal wall. If there is no disease on the vaginal wall, the conization and SLNB / RPLND is employed. If pathologic review finds no residual disease or the residual disease is more than 5 mm away from cone margin, the surgery procedure ceases; If pathologic review finds the residual disease is less than 5 mm away from cone margin, ST± upper vaginal margin resection is performed.

If the residual disease is less than 2cm in diameter, simple trachelectomy (ST) ± upper vaginal margin resection and SLNB/ RPLND is employed.

If the residual disease is greater than 2 cm and less than 4cm in diameter, radical trachelectomy (RT) and SLNB/ RPLND is employed.

If the residual disease is greater than 4 cm in diameter, fertility-sparing surgery should be abandoned.

Tow to three cycles of adjuvant chemotherapy will be administrated after the fertility-sparing surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with cervical cancer staging IB1-IIA2 desiring keeping their fertility function

Exclusion Criteria:

* retroperitoneal lymph node metastasis, involvement of lower part of uterus and endometrial carcinoma

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 5 years

SECONDARY OUTCOMES:
overall survival rate | 5years

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, PhD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Clinical Trial Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No